CLINICAL TRIAL: NCT02144506
Title: Tests and Exercises Home-based Program "T&E" for Fall Prevention and Quality of Life in Elderly: a Randomised Control Pilot-study
Brief Title: Home-based Program "T&E" for Fall Prevention and QoL in Elderly: a Randomised Control Pilot-study
Acronym: "T&E"elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HES-SO Valais-Wallis (Other)
Responsible Party: Principal Investigator, Mittaz Hager Anne-Gabrielle, Prof., HES-SO Valais-Wallis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 37715
Record Dates: First submitted 2014-05-19; First posted 2014-05-22 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Accidental Falls
Keywords: Elderly, home-based exercises programm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- T&E (Experimental): Home-based exercises program "T&E".This exercise program proposes 50 exercises with a booklet, cards and an electronic tablet. The participants choose their exercises on the basis of a rating scale of perception of exercise difficulty.
  Interventions: Other: T&E
- OTAGO (Active Comparator): Programm "OTAGO" is a home-based exercises program.
  Interventions: Other: OTAGO

INTERVENTIONS:
Other: T&E
  Other Names: Home-based exercises programm "T&E"
  Arms: T&E
Other: OTAGO
  Other Names: Home-based exercises program "OTAGO
  Arms: OTAGO

SUMMARY:
The aim of the pilot-study is to evaluate the feasability of a future RCT, regarding recruitement of eligible participants, adhesion rate, datarecording and cost. In this feasibility pilot study, 18 patients with at least 65 years will be allocated randomly to one of two interventions. The control group gets a well-known home-based exercise program (OTAGO) aiming to prevent falls where the exercises are prescribed by a physical therapists. The exercises will be presented on a booklet and on printed cards. The Intervention group consists of an exercise program, the "T&E" program, where the elderly persons can choose the exercises depending on their abilities. The exercises in the "T&E" program will be presented in a printed manual and shown on videos on an electronic tablet. Both intervention groups receive 6 hours of instruction and control/supervision sessions by physical therapists. In addition, the participants will exercise alone.

The interventions will be performed over 24 weeks.

In this pilot study, the hypothesis is that the adhesion rate is at least 65%. Other feasibility criteria will be costs, data recording issues and the qualitative evaluation of the booklet and the tablet.

Falls will be assessed with a falls calendar. The amount of physical activity of the participants is assessed with an accelerometers (actigraph) and quality of life will be assessed with OPQOL-35 at baseline, week 16 and week 24.

ELIGIBILITY:
Inclusion Criteria:

* Living at home
* Ability to perform standing position independently with/without walking aids (rollator crutch)
* Reported fall(s) during the last 12 months and/or fear of falling (Short FES-I ≥8)
* Understand french / german

Exclusion Criteria:

* Actually in treatment with a physical therapist
* Participate at an other home-based programm exercises
* MMS Score ≥ 25.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Adhesion rate | 24 weeks
  Feasability of a futur study about the recruting processus and adhesion rate (≥ 65%)

SECONDARY OUTCOMES:
Feasability | 24 weeks
  Feasability about cost, datarecording, qualitativ evaluation of the booklet and the electronic tablet

OTHER OUTCOMES:
Falls | 24 weeks
  monthly calendar
Physical activity | 24 weeks
  6 monthly calendars and accelerometer (baseline and 16st week)
Quality of life | 24 weeks
  OPQOL-35 questionnaire, at baseline, on the 16st week and end of intervention
Timed Up and Go (TUG) test | 24 weeks
  at baseline and at the end of the intervention
Functional Reach test (FR) | 24 weekds
  at baseline and at the end of the intervention
Four-Test balance scale | 24 weeks
  at the baseline and at the end of the intervention
Five Time Sit to Stand (FTSTS) | 24 weeks
  at baseline and at the end of the intervention
Walking speed | 24 weeks
  at baseline and at the end of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Anne Jacquier-Delaloye, Master, Study Director — Direction
Locations (1):
- University of Applied Sciences and Arts Western Switzerland, Sion, Valais Wallis, Switzerland